CLINICAL TRIAL: NCT00406978
Title: A Phase I/II, Multi-Center, Open Label Study of Melphalan, Prednisone, Thalidomide and Defibrotide in Advanced and Refractory Multiple Myeloma Patients
Brief Title: Melphalan, Prednisone, Thalidomide and Defibrotide in Relapsed Multiple Myeloma Patients
Acronym: MPTD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Silvio Aime (Other)
Responsible Party: Sponsor-Investigator, Silvio Aime, MD, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM2005
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Myeloma
Keywords: MYELOMA; THALIDOMIDE; DEFIBRODITE
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Prednisone; Melphalan; Thalidomide; defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MPTD (Experimental)
  Interventions: Drug: Prednisone; Drug: Melphalan; Drug: Thalidomide; Drug: Defibrotide

INTERVENTIONS:
Drug: Prednisone — Prednisone will be given orally at the dose of 1.5 mg/Kg for 4 days followed by a 31-day rest period (days 5 through 35)
Drug: Melphalan — Melphalan will be given orally at the dose of 0.25 mg/Kg for 4 days,
Drug: Thalidomide — Thalidomide will be administered orally at the initial dose of 50 mg/day p.o. once daily, with increment of 50 mg after a month to acceptable tolerance (maximum 100 mg), continuously for the entire 6 courses.
Drug: Defibrotide — Lev - 1 Def = 10 mg/Kg (max 0.6 g) on days 1-4, followed by 1.2 g (400 mg every 8 hours) p.o. through day 35 Lev - 1 Def = 1.2 g p.o (400 mg every 8 hours) on days 1-4, followed by 1.2 g (400 mg every 8 hours) p.o. through day 35 Level + 1 Def = 17 mg/Kg (max 1.2 g) on days 1-4, followed by 1.6 g p.o. (400 mg every 6 hours) through day 35 Lev + 1 Def = 2.4 g p.o. (400 mg every 4 hours) on days 1-4, followed by 1.6 g p.o. (400 mg every 6 hours) through day 35 Lev + 2 Def = 34 mg/Kg (max 2.4 g) as a i.v. injection on days 1-4, followed by 3.2 g p.o. (800 mg every 6 hours) through day 35 Lev + 2 Def = 4.8 g p.o. (800 mg every 4 hours) on days 1-4, followed by 3.2 g p.o. (800 mg every 6 hours) through day 35 Lev + 3 Def = 51mg/Kg (max 3.6 g) as a i.v. injection on days 1-4, followed by 4.8 g p.o. (1200 mg every 6 hours) through day 35 Lev + 3 Def = 7.2 g p.o.(1200 mg every 4 hours ) on days 1-4, followed by 4.8 g p.o. (1200 mg every 6 hours) given p.o. through day 35

SUMMARY:
This study will evaluate the safety and the efficacy of the association of Melphalan/ Prednisone/Thalidomide/Defibrotide (MPTD) as salvage treatment in advanced and refractory myeloma patients. This association might further increase the response rate achieved by oral MPT regimen

DETAILED DESCRIPTION:
Defibrotide (DF) is a novel orally bioavailable polydisperse oligonucleotide with anti-thrombotic and anti-adhesive effects, which has been shown to be active in various microangiopathies, including the treatment and prophylaxis of veno-occlusive disease. While DF has minimal inhibitory effect on multiple myeloma (MM) in cell isolates, it showed single agent activity on human MM xenografts in SCID/NOD mice and markedly increased responsiveness of MM to cytotoxic agents, including melphalan, cyclophosphamide and dexamethasone in the same models. DF might thus enhance the response rate of Melphalan, Prednisone and Thalidomide, while protecting against the prothrombotic state seen with this combination in the treatment of MM. In this multicenter, open label, non-randomised phase I/II trial, dosing safety and efficacy of melphalan, prednisone, thalidomide, and DF (MPTD) were determined in pts with relapsed/refractory MM.

Primary refractory or pts receiving therapeutic anticoagulation were excluded. Oral melphalan was administered at 0,25 mg/Kg on D1-4, oral prednisone at 1,5 mg/kg on D 1-4, thalidomide was delivered at 50 mg on D1-35 on cycle 1 and at 100 mg from cycle 2 to cycle 6.

Level + 1 DF = 17 mg/Kg i.v. or 2.4 g p.o. D1-4, followed by 1.6 g p.o. through D 35 Level + 2 DF = 34 mg/Kg i.v. or 4.8 g p.o. D 1-4, followed by 3.2 g p.o. through D 35 Level + 3 DF = 51 mg/Kg i.v. or 7.2 g p.o. D 1-4, followed by 4.8 g p.o. through D 35.

Each course was repeated every 35d for a total of 6 courses and no DVT prophylaxis was used.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must meet all of the following inclusion criteria to be enrolled in the study:
* Patient is of a legally consenting age as defined by local regulations.
* Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) for the duration of the study.
* Patient was previously diagnosed with multiple myeloma based on standard criteria (see Section 13.2).
* Patient is relapsed after one line of treatment but less than three lines, including high-dose chemotherapy with stem cell support, conventional poli-chemotherapy, thalidomide- and melphalan-based regimens
* Patient with primary refractory disease will be considered not eligible
* Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours.
* Patient has a Karnofsky performance status ≥60%.
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1, before study drug administration):
* Platelet count ≥90 x 109/L without transfusion support within 7 days before the test.
* Absolute neutrophil count (ANC) ≥ 1.00 x 109/L without the use of growth factors
* Corrected serum calcium ≤14 mg/dL (3.5 mmol/L).
* Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal (ULN).
* Alanine transaminase (AST): ≤ 2.5 x the ULN.
* Total bilirubin: ≤ 1.5 x the ULN.
* Calculated or measured creatinine clearance: ≥20 mL/minute

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or beast feeding females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other concomitant standard/experimental anti-myeloma drug or therapy
* Known positive for HIV or active infectious hepatitis, type B or C
* Other concurrent anticoagulation treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-02; Primary Completion 2010-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The safety will be assessed by showing DLT and maximum tolerated dose (MTD) of defibrotide when administered in combination with MPT | 7 months
  The DLT is defined by the development of febrile neutropenia, or Grade 4 neutropenia >= a week, or Grade 4 hematologic toxicity except neutropenia, or any >= Grade 3 non-hematologic toxicity considered by investigators to be related to study drug(s) in >30% of pts.
  MTD: maximum tolerated dose
The efficacy will be assessed by showing at least 55% of patients in a minimal response (MR) or at least 10 % of pts in near complete remission (nCR). | 7 months

SECONDARY OUTCOMES:
prolongation of progression-free survival | it will be evaluated from the date of enrolling until the date of first documented evidence of the end point.
duration of progression-free survival | it will be evaluated from the date of enrolling until the date of first documented evidence of the end point.
prolongs overall survival | it will be evaluated from the date of enrolling until the date of first documented evidence of the end point.

CONTACTS AND LOCATIONS:
Overall Officials: MARIO BOCCADORO, MD, Principal Investigator — DIVISIONE DI EMATOLOGIA DELL'UNIVERSITA' DI TORINO, AZIENDA OSPEDALIERA SAN GIOVANNI BATTISTA, TORINO, ITALY
Locations (5):
- Italy (5):
  - Dip. Scienze Mediche & IRCAD-Università, UDA Ematologia, Novara, Novara
  - Policlinico Monteluce, Clinica Medica I, Perugia, Perugia
  - Divisione Di Ematologia, Ospedali Riuniti, Reggio Calabria, Reggio Calabria
  - Servizio di Ematologia, Azienda Ospedaliera S. Maria Nuova, Reggio Emilia, Reggio Emilia
  - Div. Univ. Di Ematologia, Az. Osp. San Giovanni Battista, Torino, TO

REFERENCES:
- [Background] Buzaid AC, Durie BG. Management of refractory myeloma: a review. J Clin Oncol. 1988 May;6(5):889-905. doi: 10.1200/JCO.1988.6.5.889. PMID 2452861
- [Background] Palumbo A, Bertola A, Falco P, Rosato R, Cavallo F, Giaccone L, Bringhen S, Musto P, Pregno P, Caravita T, Ciccone G, Boccadoro M. Efficacy of low-dose thalidomide and dexamethasone as first salvage regimen in multiple myeloma. Hematol J. 2004;5(4):318-24. doi: 10.1038/sj.thj.6200403. PMID 15297848
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] McKean-Cowdin R, Feigelson HS, Ross RK, Pike MC, Henderson BE. Declining cancer rates in the 1990s. J Clin Oncol. 2000 Jun;18(11):2258-68. doi: 10.1200/JCO.2000.18.11.2258. PMID 10829046
- [Background] Alexanian R, Barlogie B, Tucker S. VAD-based regimens as primary treatment for multiple myeloma. Am J Hematol. 1990 Feb;33(2):86-9. doi: 10.1002/ajh.2830330203. PMID 2301376
- [Derived] Palumbo A, Larocca A, Genuardi M, Kotwica K, Gay F, Rossi D, Benevolo G, Magarotto V, Cavallo F, Bringhen S, Rus C, Masini L, Iacobelli M, Gaidano G, Mitsiades C, Anderson K, Boccadoro M, Richardson P; Italian Multiple Myeloma Network GIMEMA. Melphalan, prednisone, thalidomide and defibrotide in relapsed/refractory multiple myeloma: results of a multicenter phase I/II trial. Haematologica. 2010 Jul;95(7):1144-9. doi: 10.3324/haematol.2009.017913. Epub 2010 Jan 6. PMID 20053869